CLINICAL TRIAL: NCT06946316
Title: Dairy Versus Plant-based Beverages Combined With Resistance-training for Improving Bone Health
Brief Title: Dairy vs Plant-based Beverages for Improving Bone Health During Exercise
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 361218
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1% chocolate milk (Experimental): 375 ml of 1% chocolate milk consumed immediately after resistance training sessions + 375 ml of chocolate milk consumed 1 hour after resistance training sessions
  Interventions: Dietary Supplement: Nutritional supplementation during a 12 month resistance training program
- Pea-based beverage (Experimental): 375 ml of pea beverage consumed immediately after resistance training sessions + 375 ml of pea beverage consumed 1 hour after resistance training sessions
  Interventions: Dietary Supplement: Nutritional supplementation during a 12 month resistance training program
- Almond beverage (Placebo Comparator): 375 ml of almond beverage consumed immediately after resistance training sessions + 375 ml of almond beverage consumed 1 hour after resistance training sessions
  Interventions: Dietary Supplement: Nutritional supplementation during a 12 month resistance training program

INTERVENTIONS:
Dietary Supplement: Nutritional supplementation during a 12 month resistance training program — 1% chocolate milk
  Arms: 1% chocolate milk
Dietary Supplement: Nutritional supplementation during a 12 month resistance training program — pea-based beverage
  Arms: Pea-based beverage
Dietary Supplement: Nutritional supplementation during a 12 month resistance training program — almond-based beverage
  Arms: Almond beverage

SUMMARY:
This study will evaluate the effects of consuming dairy milk versus two plant-based beverages (pea-based, and almond-based) after resistance training sessions (3 times per week for 12 months) on bone properties (bone mineral density, bone geometry), body composition, strength, and functional performance in post-menopausal women and men 50y and older.

DETAILED DESCRIPTION:
The purpose of the study is to compare consumption of dairy milk (1% chocolate milk) to plant-based beverages (protein-matched pea beverage and low-protein almond beverage) after resistance-training sessions on bone mineral density, bone geometric properties, lean tissue and fat mass, muscular strength, and functional performance. One-hundred and fifty postmenopausal women and men 50y or older will be randomized to one of three groups: 1) Dairy milk; 2) pea-beverage; 3) almond beverage. The study will be double-blind, accomplished by chocolate flavoring of each beverage. Participants will do supervised strength-training sessions three times per week for 12 months. After each strength-training session, participants will consume 375 ml of their beverage and then consume 375 ml of their beverage again one hour later.

ELIGIBILITY:
Inclusion Criteria:

* Women need to be postmenopausal (no age limit)
* Men need to be 50y or older

Exclusion Criteria:

* Taking medications that might affect bone
* Conditions that might preclude participating in a resistance-training program (determined by the "Get Active Questionnaire").
* Planning 6 weeks of travel during the 12 month intervention period
* Planning major surgery during the 12 month intervention period
* Already strength training greater than 2 days per week for 30 minutes or longer per session
* Allergies to ingredients in the beverages

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in section modulus at the hip (cm to the power of 3) | 12 months
  Section modulus measured by dual energy X-ray absorptiometry

SECONDARY OUTCOMES:
Change in lumbar spine bone mineral density (g/cm-squared) | 12 months
  Lumbar spine bone mineral density measured by dual energy X-ray absorptiometry
Change in hip bone mineral density (g/cm-squared) | 12 months
  Hip bone mineral density measured by dual energy X-ray absorptiometry
Change in cross-sectional area at the hip (cm-squared) | 12 months
  Cross-sectional area measured by dual energy X-ray absorptiometry
Change in cortical thickness at the hip (cm) | 12 months
  Cortical thickness measured by dual energy X-ray absorptiometry
Change in buckling ratio at the hip (no units) | 12 months
  Buckling ratio measured by dual energy X-ray absorptiometry
Change in bench press strength (kg) | 6 and 12 months
  Bench press strength determine from 1-repetition maximum
Change in knee extension strength (kg) | 6 and 12 months
  Knee extension strength determined from 1-repetition maxium
Change in lean tissue mass (kg) | 12 months
  Lean tissue mass measured by dual energy X-ray absorptiometry
Change in fat mass (kg) | 12 months
  Fat mass measured by dual energy X-ray absorptiometry
change in 30 second sit to stand (number of repetitions) | 6 and 12 months
  Maximal number of times sitting and standing in 30 seconds
Change in walking speed (m/s) | 6 and 12 months
  walking speed measured over 10 m
Change in timed up and go performance (s) | 6 and 12 months
  Time for standing from a chair, walking 6 meters and sitting back down

CONTACTS AND LOCATIONS:
Locations (1):
- College of Kinesiology University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No